CLINICAL TRIAL: NCT01241851
Title: Effect of Acute Exercise on Cognitive Functions
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: The Zinman College for Physical Education and Sport Exercise, Wingate Institute (Unknown)
Responsible Party: Prof. R. Caraso, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Single Group | Purpose: Prevention
Other Study IDs: 0093-10-HYMC
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Cognitive Function in Elderly
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aerobic exercise (Active Comparator)
  Interventions: Behavioral: Aerobic exercise
- Resistance exercise (Active Comparator)
  Interventions: Behavioral: Resistance exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Aerobic exercise
  Arms: Aerobic exercise
Behavioral: Resistance exercise
  Arms: Resistance exercise

SUMMARY:
To determine whether acute aerobic exercise versus resistance exercise effects cognitive function among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Exercise at least 2 times a week Able to sign informed consent Able to perform ergometric exam Above 40 years old

Exclusion Criteria:

* Smoking
* Suffering psychiatric or neurologic illness
* No medication for chronic illness that could effect cognitive function
* Problems with cognitive functioning after head trauma
* Long-term hospitalization within the past 3 months
* Inability to use computer because of vision or motor problems
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Level of executive function | One month

CONTACTS AND LOCATIONS:
Locations (1):
- Zinman College, Wingate Institute, Netanya, Israel